CLINICAL TRIAL: NCT01051024
Title: Efficacy of Diamel in the Treatment of Polycystic Ovary Syndrome
Brief Title: Diamel in the Treatment of Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-0917-CU
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Dietary supplement; Diamel; Polycystic Ovary Syndrome; Female Infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Diamel
  Interventions: Dietary Supplement: Diamel
- B (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Diamel — Two Diamel tablets (Orally administered) three times a day (just before each meal: breakfast, lunch and dinner), for 24 weeks.
  Arms: A
Dietary Supplement: Placebo — Two Placebo tablets (Orally administered) three times a day (just before each meal: breakfast, lunch and dinner), for 24 weeks.
  Arms: B

SUMMARY:
The purpose of this study is to assess the efficacy of Diamel administration in the treatment of Polycystic Ovary Syndrome. The duration of this double-blind placebo controlled phase 3 clinical trial will be 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Two of the following criteria:

  * Oligo or Anovulation
  * Polycystic Ovary diagnosed by ultrasound technique
  * Clinical signs of Hyperandrogenism
* Signed informed consent

Exclusion Criteria:

* Personal history of other causes of hyperandrogenism: Hyperprolactinemia, suprarenal tumors, ovary tumors, suprarenal hyperplasia, hypercortisolism.
* Patients under other experimental treatment
* Treatment with ovulation inducers and/or insulin sensitizers within 60 days before treatment
* Treatment with vitamins within 7 days before treatment
* Treatment with dietary supplements within 60 days before treatment
* Non-compensated intercurrent diseases: diabetes mellitus, thyroid disease, hypertension

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Normalization of blood concentrations of androgens at week 24 | 24 weeks
Normalization of blood concentrations prolactin at week 24 | 24 weeks
Normalization of blood concentrations of estrogens at week 24 | 24 weeks
Normalization of blood concentrations of FSH at week 24 | 24 weeks
Normalization of blood concentrations of LH at week 24 | 24 weeks

SECONDARY OUTCOMES:
Regularization of the menstrual cycle at week 24. | 24 weeks
Reappearance of ovulatory cycles at week 24 | 24 weeks
Normalization of blood concentrations of insulin at week 24 | 24 weeks
Normalization of blood concentrations of cholesterol at week 24 | 24 weeks
Normalization of blood concentrations of triglycerides at week 24 | 24 weeks
Normalization of blood concentrations of glucose at week 24 | 24 weeks
Improvement of clinical signs associated with polycystic ovary syndrome: acne, hirsutism, abdominal obesity, and blood pressure at week 24. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Hernandez, MD, Principal Investigator — "Ramón González Coro" Gynecologic and Obstetric Hospital
Locations (1):
- "Ramón González Coro" Gynecologic and Obstetric Hospital, Havana, La Habana, Cuba